CLINICAL TRIAL: NCT04642937
Title: Study of CD200 Activation Receptor Ligand (CD200AR-L) and Allogeneic Tumor Lysate Vaccine Immunotherapy for Recurrent Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OX2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRPC #2017LS096
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hP1A8 (Experimental): Up to 3 dose levels of hP1A8 will be tested with a Dose Level -1 in the event of toxicity. The MTD will be identified using the standard 3+3 design. Upon determination of the MTD, additional patients will be enrolled as part of an expansion cohort.
  Interventions: Drug: Treatment with hP1A8

INTERVENTIONS:
Drug: Treatment with hP1A8 — Treatment with hP1A8

SUMMARY:
This is a single-center, open-label, dose-range finding Phase I study of hP1A8, a new adjuvant CD200 activation receptor ligand (CD200AR-L), in combination with imiquimod and the GBM6-AD vaccine to treat recurrent glioblastoma (GBM) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older.
* Confirmed diagnosis of GBM.
* Radiographically or histologically proven progression or recurrence of disease at any time after standard of care therapy (radiation, temozolomide, with or without a tumor treatment field device).
* Tumor debulking or biopsies may be performed to clinical trial enrollment if indicated and feasible.

Exclusion Criteria:

* Bevacizumab or targeted therapy within 45 days of enrollment.
* Intercurrent immune system disorder such as hypoimmunity (marrow failure, HIV) or hyperimmunity (autoimmune disease).
* Unable to complete a standard upfront course of chemoradiotherapy due to disease progression or intolerance of therapy.
* History of Gliadel water, GammaTile or other implanted therapeutic agent.
* Concurrent use of tumor treatment field devices (e.g. Optune).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of hP1A8 when administered with imiquimod and GBM6-AD | 12 months

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) | 12 months
Time to progression (TTP) | 24 months
Progression free survival (PFS) | 24 months
Overall survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States